CLINICAL TRIAL: NCT04528732
Title: Suubi4Stigma: Addressing HIV-Associated Stigma Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH121141 (NIH)
Record Dates: First submitted 2020-08-03; First posted 2020-08-27 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: Adolescents will be randomly assigned to one of three study arms: 1) Usual care to receive the currently implemented usual care addressing HIV/AIDS-associated stigma (educational materials from the Ugandan Ministry of Health); 2) G-CBT intervention + Usual care; and 3) MFG intervention + Usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Usual care consists of the traditional clinic intervention that focuses on testing services, ART treatment, and information about disease management.
- Group-Cognitive Behavioral Therapy (G-CBT) (Experimental): G-CBT consists of 10-session for HIV/AIDS-associated stigma, utilizing core components of CBT, including psychoeducation, cognitive restructuring, and skill-building to increase adaptive coping mechanisms.
  Interventions: Behavioral: Group Cognitive Behavioral Therapy (G-CBT)
- Multiple Family Group (MFG) (Experimental): MFG consists of 10-sessions that strengthen family relationships intended to address HIV/AIDS-associated stigma at the individual level and within families. The core components of MFG are known as 4Rs and 2S's: rules, responsibility, relationships, respectful communication, stress and social support.
  Interventions: Behavioral: Multiple Family Group (MFG)

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy (G-CBT) — G-CBT consists of 10-session for HIV/AIDS-associated stigma, utilizing core components of CBT, including psychoeducation, cognitive restructuring, and skill-building to increase adaptive coping mechanisms.
  Arms: Group-Cognitive Behavioral Therapy (G-CBT)
Behavioral: Multiple Family Group (MFG) — MFG consists of 10-sessions that strengthen family relationships intended to address HIV/AIDS-associated stigma at the individual level and within families. The core components of MFG are known as 4Rs and 2S's: rules, responsibility, relationships, respectful communication, stress and social support.
  Arms: Multiple Family Group (MFG)

SUMMARY:
The study seeks to reduce HIV/AIDS-associated stigma and its negative impact on adolescent health and psychosocial well-being. This study will examine two evidence-informed interventions: 1) group cognitive behavior therapy (G-CBT) that aims at cognitive restructuring and strengthening coping skills at the individual level, and 2) multiple family group (MFG) that strengthens family relationships intended to address HIV/AIDS-associated stigma at the individual level and within families. Adolescents between 10-14 years, will be randomly assigned -at the clinic level, to one of three study arms: 1) Usual care to receive the currently implemented usual care addressing HIV/AIDS-associated stigma (educational materials from the Ugandan Ministry of Health); 2) G-CBT intervention + Usual care; and 3) MFG intervention + Usual care. The interventions will be delivered over a 3-month period. Assessments will be collected at baseline, 3 months and 6 months post intervention initiation. The study will also explore participants, caregivers and facilitators' intervention experiences, as well as multi-level facilitators and barriers to intervention implementation and participation.

DETAILED DESCRIPTION:
Sub-Saharan Africa (SSA) is heavily burdened by HIV, with 85% of new infections among adolescents and youth globally happening in the region. Recent statistics indicate that HIV prevalence among adolescents and young people is rising in Uganda. While availability and access to free antiretroviral therapy (ART) has decreased child mortality, it has increased the likelihood that a number of children living with HIV (CLWH) will transition into adulthood, with HIV as a chronic, highly stigmatized illness. Unfortunately, the stigma this group experiences results in much lower quality of life. Stigma, a common experience characterized by public blame, moral condemnation and discrimination, has been documented to be one of the greatest challenges to slowing the spread of HIV&AIDS. It perpetuates the culture of silence and fear and prevents individuals from testing and seeking health care. Research has shown that HIV/AIDS-associated stigma predicts depression and PTSD, poor treatment and adherence, loneliness and social isolation, HIV-related physical health, and HIV sexual risk behavior. It is critical for HIV interventions to target stigma in order to reduce HIV spread. Yet, stigma-reduction interventions targeting children and adolescents living with HIV/AIDS in SSA are almost non-existent. Thus, there is a need for research that will generate knowledge to address HIV/AIDS-associated stigma, especially among CLWH as they transition to adolescence. The proposed exploratory study (R21) will: Aim 1: Pilot test the feasibility, acceptability, and preliminary impact of an innovative Group Cognitive Behavior Therapy (G-CBT) and Multiple Family Group (MFG) interventions on reducing HIV/AIDS-associated stigma and its impact on targeted participant outcomes (stigma, post-trauma symptoms, depression, sexual risk behavior, family/social support, and adherence to medication) in comparison to: 1a) usual care vs G-CBT; 1b) Usual care vs MFG; 1c) G-CBT vs. MFG. Aim 2: Qualitatively examine participants' and facilitators' intervention experiences and identify individual, family and institutional-level facilitators and barriers to G-CBT and MFG intervention implementation and participation. The study will be conducted in 9 health clinics (n = 90 children, ages 10-14) and their caregivers (total 90 child- caregiver dyads) in Masaka. Clinics will be randomized to one of three study arms (n=3 clinics; 30 child-caregiver dyads each arm): 1) Usual care to receive the currently implemented usual care addressing HIV/AIDS-associated stigma (educational materials developed by the Ugandan Ministry of Health); 2) G-CBT intervention + usual care; and 3) MFG intervention + usual care. Participants will be followed over a 6-month period, with data collected at baseline, 3 months and 6 months post intervention initiation to assess feasibility, acceptability, and preliminary impact. The long-term goal of the proposed research is to develop culturally appropriate, feasible, acceptable and effective interventions that address HIV/AIDS-associated stigma and its impact on CLWH's wellbeing and their families in SSA.

ELIGIBILITY:
Inclusion Criteria for Children:

1. HIV+ status - defined as a child who has been tested for HIV with confirmation by medical report and has been disclosed to, i.e. know their status
2. Prescribed antiretroviral therapy
3. Living within a family (defined broadly - not necessarily with biological parents)
4. Ages 10 to 14 years.

   Exclusion Criteria for Children:
5. Unable to understand the study procedures and/or participant rights during the informed consent process
6. Unwilling or unable to commit to completing the study.
7. Presents with emergency needs (e.g., hospitalization), needed care will be secured, rather than study participation

Inclusion Criteria for Caregivers:

1. Ages 18 and above
2. Agree to participate in the study.

   Exclusion Criteria for Caregivers
3. Unable to understand the study procedures and/or participant rights during the informed consent process
4. Unwilling or unable to commit to completing the study.
5. Presents with emergency needs (e.g., hospitalization), needed care will be secured, rather than study participation

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Washington University in St. Louis, St Louis, Missouri, United States
- Uganda (2):
  - International Center for Child Health and Development Field Office, Masaka
  - Reach the Youth Uganda, Masaka

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PI and indicates the data will be used for the purposes of research (per Code of Federal Regulations Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Washington University in St. Louis' Office of Sponsored Projects' data sharing agreement.
Supporting Information: Analytic Code

REFERENCES:
- [Derived] Nabunya P, Ssewamala FM, Kizito S, Mugisha J, Brathwaite R, Neilands TB, Migadde H, Namuwonge F, Ssentumbwe V, Najjuuko C, Sensoy Bahar O, Mwebembezi A, McKay MM. Preliminary Impact of Group-Based Interventions on Stigma, Mental Health, and Treatment Adherence Among Adolescents Living with Human Immunodeficiency Virus in Uganda. J Pediatr. 2024 Jun;269:113983. doi: 10.1016/j.jpeds.2024.113983. Epub 2024 Feb 23. PMID 38401789
- [Derived] Kizito S, Nabunya P, Ssewamala FM. Enhancing Adherence to Antiretroviral Therapy Among Adolescents Living With HIV Through Group-Based Therapeutic Approaches in Uganda: Findings From a Pilot Cluster-Randomized Controlled Trial. J Pediatr Psychol. 2023 Nov 16;48(11):907-913. doi: 10.1093/jpepsy/jsad081. PMID 37935531
- [Derived] Nabunya P, Namuwonge F, Sensoy Bahar O, Ssentumbwe V, Migadde H, Mugisha J, Ssewamala FM. Stigma by Association, Parenting Stress, and the Mental Health of Caregivers of Adolescents Living With HIV in Uganda. J Adolesc Health. 2023 May;72(5S):S18-S23. doi: 10.1016/j.jadohealth.2022.08.017. PMID 37062579
- [Derived] Nabunya P, Ssewamala FM, Bahar OS, Michalopoulos LTM, Mugisha J, Neilands TB, Trani JF, McKay MM. Suubi4Stigma study protocol: a pilot cluster randomized controlled trial to address HIV-associated stigma among adolescents living with HIV in Uganda. Pilot Feasibility Stud. 2022 Apr 29;8(1):95. doi: 10.1186/s40814-022-01055-7. PMID 35488323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited children and their caregivers (dyads). A total of 89 dyads (N=178) were recruited from 9 health clinics. Dyads were randomized (at the clinic level) to three study groups: Usual care (n=29 dyads), MFG-FS (n=34 dyads) and G-CBT (n=26 dyads).
Period: Overall Study
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Started (child-caregiver dyads) | 29 | 26 | 34
Completed (child-caregiver dyads) | 28 | 25 | 31
Not Completed | 1 | 1 | 3
Not completed — Death | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The study recruited a total of 89 child and their caregivers (N=89 dyads). The total number of participants (both children and caregivers) is N=178. Baseline measures were analyzed separately for children and caregivers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG) | Total
Number analyzed (Participants) | 58 | 52 | 68 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] — The study recruited both children and their caregivers (n=89 dyads). Total includes both children and caregivers. Population: Age was analyzed separately for children and caregivers.
  years
    Child age: number analyzed (Participants) | 29 | 26 | 34 | 89
    Child age | 12.45 (1.35) | 12.69 (1.09) | 11.65 (1.52) | 12.21 (1.41)
    Caregiver age: number analyzed (Participants) | 29 | 26 | 34 | 89
    Caregiver age | 48.69 (13.40) | 46.77 (11.22) | 46.65 (16.77) | 47.35 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants] — The study recruited both children and their caregivers (n=89 dyads). Total includes both children and caregivers. Population: Sex was analysed separately for children and caregivers.
  Participants
    Child Sex: number analyzed (Participants) | 29 | 26 | 34 | 89
    Child Sex: Female | 17 | 17 | 22 | 56
    Child Sex: Male | 12 | 9 | 12 | 33
    Caregiver sex: number analyzed (Participants) | 29 | 26 | 34 | 89
    Caregiver sex: Female | 22 | 18 | 29 | 69
    Caregiver sex: Male | 7 | 8 | 5 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was analyzed separately for children and caregivers.
  Participants
    Child Race: number analyzed (Participants) | 29 | 26 | 34 | 89
    Child Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Child Race: Asian | 0 | 0 | 0 | 0
    Child Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Child Race: Black or African American | 29 | 26 | 34 | 89
    Child Race: White | 0 | 0 | 0 | 0
    Child Race: More than one race | 0 | 0 | 0 | 0
    Child Race: Unknown or Not Reported | 0 | 0 | 0 | 0
    Caregiver Race: number analyzed (Participants) | 29 | 26 | 34 | 89
    Caregiver Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Caregiver Race: Asian | 0 | 0 | 0 | 0
    Caregiver Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Caregiver Race: Black or African American | 29 | 26 | 34 | 89
    Caregiver Race: White | 0 | 0 | 0 | 0
    Caregiver Race: More than one race | 0 | 0 | 0 | 0
    Caregiver Race: Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Child and Caregiver Region on enrollment (N= 89 child-caregiver dyads). Number of children = 89; number of caregivers = 89
  Participants
    Uganda: Children | 29 | 26 | 34 | 89
    Uganda: Caregivers | 29 | 26 | 34 | 89
HIV Stigma (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Child HIV Stigma was measured by the HIV Stigma Scale (HSS). The 40-item scale measures stigma and psychosocial aspects of having HIV. Responses were rated on a 4-point scale with 1= strongly agree, 2= agree, 3=disagree and 4=strongly disagree. Items in the inverse direction were reverse coded to create summated scores, with higher scores indicating high levels of HIV-related stigma. The theoretical range for this scale is 40-160. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 84.41 (19.60) | 79.15 (19.25) | 77.88 (18.74) | 80.38 (19.17)
HIV Shame (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Child HIV Shame was measured by the Shame Questionnaire. The 8-item scale is used to assess child's feelings of shame on a 3-point scale, with 0 =not true, 1 = somewhat true and 2 =very true. Summated scores were created with higher scores representing high levels of HIV-associated shame. The theoretical range is 0-16. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 3.28 (3.78) | 2.54 (2.34) | 2.59 (2.87) | 2.80 (3.05)
Stigma by Association (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Stigma by association (Child reports) was measured using 10-items from the Brief Stigma-by Association Scale. The scale measures experiences and consequences of associated stigma, on a 3-point scale with 0= Not at all, 1= Sometimes and 2= All the time. Summated scores were created with higher scores indicating high levels of stigma-by association. The theoretical range for the scale is 0-20. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 4.38 (4.76) | 4.73 (5.14) | 2.88 (3.78) | 3.91 (4.56)
Depressive Symptoms (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — The Child Depression Inventory (CDI) was used to measure children's depressive symptoms. Respondents were asked to mark a statement that best described their feelings during the past 2 weeks. Each of the 14-items on the CDI has three response options that correspond to varying levels of symptomology for clinical depression. The theoretical range for this scale is 0-28, with higher scores representing high levels of depressive symptoms. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 4.90 (3.48) | 5.38 (3.49) | 4.85 (3.82) | 5.02 (3.58)
Self-Concept (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Self-concept was measured using the Tennessee Self-Concept Scale (TSCS). The 20-item scale measures children's perception of identity, self-satisfaction and other behaviors. Each item was rated on a 5-point scale: 1= always false, 2=usually false, 3=sometimes true/sometimes false, 4=usually true and 5= always true (theoretical range: 20-100). Ten items in the inverse direction were reverse coded to create summated scores, with higher scores indicating higher levels of child self-concept. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 38.03 (5.80) | 39.92 (7.53) | 36.39 (7.41) | 38.01 (7.01)
Hopelessness (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Hopelessness was measured using the Beck Hopelessness Scale (BHS). The 20-item scale measures children's hopelessness and pessimistic attitudes toward the future. Items have a "true" or "false" response coded as "1" or "0" respectively. Nine items with positive wording were reverse coded to create a summated score for the entire scale. The theoretical range for the BHS is 0-20, with higher scores indicating higher levels of hopelessness. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 6.00 (3.22) | 6.27 (3.42) | 5.50 (3.03) | 5.89 (3.19)
Post-Traumatic Stress Disorder Symptoms (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Child PTSD was measured using 31 items from the abbreviated Childhood post-traumatic Stress Reaction Index (CPTS-RI). Participants were asked about reactions people sometimes have after very bad things happen and how this was applicable to them in the past month. Responses were rated on a 5-point Likert scale, with 0= None, 1= Little (1-2 days a week), 2 = some (2-3 days a week), 3 =Much (2 days a month) and 4 =most (Almost every day). The theoretical range is 0-124. Summated scores were created with higher scores indicating higher levels of child PTSD symptoms. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 19.76 (3.25) | 22.88 (15.69) | 20.56 (4.94) | 20.98 (14.53)
Self reported medication adherence (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Child self-reported adherence was assessed using three items: 1) "In the last 30 days, on how many days did you miss at least one dose of your HIV medications (range: 0-30 days)?" 2) "In the last 30 days, how often did you take your HIV medicine in the way you were supposed to (never to always)?" and 3) "In the last 30 days, how good a job did you do at taking your HIV medicine in the way you were supposed to (very poor - excellent)"? Responses were linearized into a continuous scale ranging from 0-100, with low scores representing poor adherence and 100 representing perfect adherence. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 90.15 (12.17) | 91.77 (9.82) | 92.55 (9.31) | 91.77 (9.82)
Engagement in sexual risk behavior (Child Reports) [Count of Participants; unit: Participants] — Engagement in sexual risk behaviors was measured by asking a respondent whether they had engaged in unprotected sex, coded as "yes" or "no". Population: Only child reports were analyzed.
  Participants
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 1 | 0 | 0 | 1
Intentions to engage in sexual risk behaviors (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Intentions to engage in sexual risk behaviors were assessed by asking respondents to rate how 5 sexual activity-related statements applied to them. Items were rated on a 5-point Likert scale, with 1=never, 2=sometimes, 3=about half of the time, 4=most of the time and 5=always. The theoretical range for this scale is 5-25, with higher scores indicating high intentions to engage in sexual risk-taking behaviors. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 6.52 (2.46) | 5.85 (2.41) | 5.91 (2.01) | 6.09 (2.27)
Child-Caregiver Support (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Child-caregiver support was measured using 17 items from the Social Support Behaviors Scale (SS-BS) scale. Respondents were asked to rate the adults they live with, on a 5-point Likert scale, with 1= never, 2 = sometimes, 3=about half of the time, 4=most of the time, and 5= always. The theoretical range for this scale is 17-85. Summated scores were created with high scores indicating high levels of perceived support from caregivers Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 54.59 (4.44) | 54.08 (5.89) | 57.00 (6.81) | 55.30 (5.89)
Friendship Quality (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Child's quality of friendships was measured using 21-items from the Friendship Qualities Scale. This multidimensional measurement scale assesses the quality of children's relationships with their best friends via several aspects, including closeness, help, safety and closeness. Respondents were asked to rate how each statement applied to them. Responses were rated on a 5- point Likert scale, with 1=never, 2=sometimes, 3=about half of the time, 4=most of the time, and 5= always. The theoretical range for this scale is 21-105, with high scores indicating high quality friendship levels. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 74.34 (15.16) | 79.08 (13.40) | 80.61 (16.67) | 78.03 (15.30)
Loneliness (Child Reports) [Mean (Standard Deviation); unit: score on a scale] — Child loneliness was assessed using the UCLA Loneliness Scale. The 20-item scale measures one's subjective feelings of loneliness as well as feelings of social isolation. Responses were rated on 4-point Likert scale with 3= I often feel this way, 2= I sometimes feel this way, 1 = I rarely feel this way, and 0=I never feel this way. The theoretical range for this scale is 0-60, with high scores indicating higher levels of social isolation. Population: Only child reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 34 (10.80) | 32.23 (11.67) | 33.47 (10.28) | 33.28 (10.77)
Stigma by Association (Caregiver Reports) [Mean (Standard Deviation); unit: score on a scale] — Stigma by association was measured using 10-items from the Brief Stigma-by-Association Scale. The scale measures experiences and consequences of associated stigma, on a 3-point scale, with 0= Not at all, 1= Sometimes and 2= All the time. The theoretical range for the scale is 0-20. Summated scores were created with higher scores indicating higher levels of stigma by association experienced by caregivers. Population: Only caregiver reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 4.90 (5.17) | 4.23 (4.85) | 5.00 (5.52) | 4.74 (5.17)
HIV/AIDS Stigma and Discrimination (Caregiver Reports) [Mean (Standard Deviation); unit: score on a scale] — The HIV/AIDS Stigma and Discrimination Scale was used. The 22-item scale assessed respondents about what they think about people living with HIV/AIDS. Responses were rated on a 4-point scale with 1= strongly agree, 2= agree, 3=disagree and 4=strongly disagree. The theoretical range for this scale is 22- 88, with higher scores indicating higher levels of perceived HIV-related stigma and discriminatory attitudes among caregivers. Population: Only caregiver reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 42.72 (9.95) | 38.85 (11.90) | 36.50 (10.51) | 39.21 (10.96)
Caregiver Mental Health (Caregiver Reports) [Mean (Standard Deviation); unit: score on a scale] — Caregiver mental health functioning was assessed using 34-items from the Brief Symptom Inventory (BSI). The scale measures symptoms of anxiety, somatization and depression. Respondents were asked to rate how they felt emotionally, on a 5-point Likert scale, with 1=Never true, 2=rarely true, 3= true sometimes, 4= true most of the time and 5=always true. The theoretical range for this scale is 34-170, with higher scores representing higher levels of caregiver mental distress. Population: Only caregiver reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 76.28 (24.36) | 75.54 (23.76) | 72.29 (20.00) | 74.54 (22.42)
Parenting Stress (Caregiver Reports) [Mean (Standard Deviation); unit: score on a scale] — Parenting stress was measured by 33 items from the Parenting Stress Index (PSI). The 33-item scale assesses symptoms related to parental distress, difficult child, and caregiver-child dysfunctional relationships. Respondents were asked to rate their parenting stress, on a 4-point Likert scale, with 1=strongly disagree, 2=somewhat disagree, 3=somewhat agree and 4=strongly agree. The theoretical range for this scale is 33-132, with high scores indicating high levels of parenting stress. Population: Only caregiver reports were analyzed.
  score on a scale
    number analyzed (Participants) | 29 | 26 | 34 | 89
    (all) | 71.17 (17.32) | 75.65 (19.93) | 70.26 (17.53) | 72.13 (18.14)

OUTCOME MEASURES:

1. Primary Outcome: HIV Stigma (Child Reports)
Description: Child HIV Stigma was measured by the HIV Stigma Scale (HSS). The 40-item scale measures stigma and psychosocial aspects of having HIV. Responses were rated on a 4-point scale with 1= strongly agree, 2= agree, 3=disagree and 4=strongly disagree. Items in the inverse direction were reverse coded to create summated scores, with higher scores indicating high levels of HIV-related stigma. Min/max values: 40-160. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 75.07 (15.35) | 73.0 (16.90) | 75.29 (18.77)

2. Primary Outcome: HIV Shame (Child Reports)
Description: Child HIV Shame was measured by the Shame Questionnaire. The 8-item scale is used to assess child's feelings of shame on a 3-point scale, with 0 =not true, 1 = somewhat true and 2 =very true. Summated scores were created with higher scores representing high levels of HIV-associated shame. Min/max values: 0-16. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 0.72 (1.44) | 0.48 (1.12) | 0.82 (1.15)

3. Primary Outcome: Stigma by Association (Child Reports)
Description: Stigma by association (Child reports) was measured using 10-items from the Brief Stigma-by Association Scale. The scale measures experiences and consequences of associated stigma, on a 3-point scale with 0= Not at all, 1= Sometimes and 2= All the time. Summated scores were created with higher scores indicating high levels of stigma-by association. Min/max values: 0-20. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 0.43 (0.74) | 1.44 (2.99) | 1.74 (3.04)

4. Primary Outcome: HIV/AIDS Stigma and Discrimination (Caregiver Reports)
Description: The HIV/AIDS Stigma and Discrimination Scale was used. The 22-item scale assessed respondents about what they think about people living with HIV/AIDS. Responses were rated on a 4-point scale with 1= strongly agree, 2= agree, 3=disagree and 4=strongly disagree. Min/max values: 22- 88, with higher scores indicating higher levels of perceived HIV-related stigma and discriminatory attitudes among caregivers. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only caregiver reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 37.36 (10.80) | 30.68 (8.88) | 33.52 (8.90)

5. Primary Outcome: Stigma by Association (Caregiver Reports)
Description: Stigma by association was measured using 10-items from the Brief Stigma-by-Association Scale. The scale measures experiences and consequences of associated stigma, on a 3-point scale, with 0= Not at all, 1= Sometimes and 2= All the time. Min/max values: 0-20. Summated scores were created with higher scores indicating higher levels of stigma by association experienced by caregivers. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only caregiver reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 3.43 (4.50) | 3.20 (4.34) | 2.58 (3.80)

6. Secondary Outcome: Child Depressive Symptoms (Child Reports)
Description: The Child Depression Inventory (CDI) was used to measure children's depressive symptoms. Respondents were asked to mark a statement that best described their feelings during the past 2 weeks. Each of the 14-items on the CDI has three response options that correspond to varying levels of symptomology for clinical depression. Min/max: 0-28, with higher scores representing high levels of depressive symptoms. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 3.28 (2.07) | 3.10 (2.57) | 4.18 (3.33)

7. Secondary Outcome: Self-Concept (Child Reports)
Description: Self-concept was measured using the Tennessee Self-Concept Scale (TSCS). The 20-item scale measures children's perception of identity, self-satisfaction and other behaviors. Each item was rated on a 5-point scale: 1= always false, 2=usually false, 3=sometimes true/sometimes false, 4=usually true and 5= always true. Min/max values: 20-100. Ten items in the inverse direction were reverse coded to create summated scores, with higher scores indicating higher levels of child self-concept. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 38.28 (4.96) | 34.61 (7.04) | 37.39 (6.18)

8. Secondary Outcome: Hopelessness (Child Reports)
Description: Hopelessness was measured using the Beck Hopelessness Scale (BHS). The 20-item scale measures children's hopelessness and pessimistic attitudes toward the future. Items have a "true" or "false" response coded as "1" or "0" respectively. Nine items with positive wording were reverse coded to create a summated score for the entire scale. Min/max values: 0-20, with higher scores indicating higher levels of hopelessness. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 4.14 (2.90) | 4.55 (3.30) | 5.00 (3.87)

9. Secondary Outcome: Post-Traumatic Stress Disorder Symptoms (Child Reports)
Description: Child PTSD was measured using 31 items from the abbreviated Childhood post-traumatic Stress Reaction Index (CPTS-RI). Participants were asked about reactions people sometimes have after very bad things happen and how this was applicable to them in the past month. Responses were rated on a 5-point Likert scale, with 0= None, 1= Little (1-2 days a week), 2 = some (2-3 days a week), 3 =Much (2 days a month) and 4 =most (Almost every day). Min/max values: 0-124. Summated scores were created with higher scores indicating higher levels of child PTSD symptoms. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 12.21 (12.47) | 9.24 (10.91) | 13.06 (12.84)

10. Secondary Outcome: Self-Reported Medication Adherence (Child Reports)
Description: Child self-reported adherence was assessed using three items: 1) "In the last 30 days, on how many days did you miss at least one dose of your HIV medications (range: 0-30 days)?" 2) "In the last 30 days, how often did you take your HIV medicine in the way you were supposed to (never to always)?" and 3) "In the last 30 days, how good a job did you do at taking your HIV medicine in the way you were supposed to (very poor - excellent)"? Responses were linearized into a continuous scale ranging from 0-100, with low scores representing poor adherence and 100 representing perfect adherence. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 93.14 (9.24) | 88.41 (15.30) | 91.37 (9.59)

11. Secondary Outcome: Engagement in Sexual Risk Behaviors (Child Reports)
Description: Engagement in sexual risk behaviors was measured by asking a respondent whether they had engaged in unprotected sex, coded as "yes" or "no". Number of participants who responded "yes" at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
Participants | 0 | 0 | 0

12. Secondary Outcome: Intentions to Engage in Sexual Risk Behaviors (Child Reports)
Description: Intentions to engage in sexual risk behaviors were assessed by asking respondents to rate how 5 sexual activity-related statements applied to them. Items were rated on a 5-point Likert scale, with 1=never, 2=sometimes, 3=about half of the time, 4=most of the time and 5=always. Min/max values: 5-25, with higher scores indicating high intentions to engage in sexual risk-taking behaviors. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 5.43 (0.92) | 5.84 (1.84) | 5.52 (1.55)

13. Secondary Outcome: Child-Caregiver Support (Child Reports)
Description: Child-caregiver support was measured using 17 items from the Social Support Behaviors Scale (SS-BS) scale. Respondents were asked to rate the adults they live with, on a 5-point Likert scale, with 1= never, 2 = sometimes, 3=about half of the time, 4=most of the time, and 5= always. Min/max values: 17-85. Summated scores were created with high scores indicating high levels of perceived support from caregivers. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 57.93 (5.91) | 54.82 (6.89) | 59.77 (5.32)

14. Secondary Outcome: Friendship Quality (Child Reports)
Description: Child's quality of friendships was measured using 21-items from the Friendship Qualities Scale. This multidimensional measurement scale assesses the quality of children's relationships with their best friends via several aspects, including closeness, help, safety and closeness. Respondents were asked to rate how each statement applied to them. Responses were rated on a 5- point Likert scale, with 1=never, 2=sometimes, 3=about half of the time, 4=most of the time, and 5= always. Min/max values: 21-105, with high scores indicating high quality friendship levels. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 78.21 (12.31) | 83.45 (15.02) | 80.50 (15.07)

15. Secondary Outcome: Loneliness (Child Reports)
Description: Child loneliness was assessed using the UCLA Loneliness Scale. The 20-item scale measures one's subjective feelings of loneliness as well as feelings of social isolation. Responses were rated on 4-point Likert scale with 3= I often feel this way, 2= I sometimes feel this way, 1 = I rarely feel this way, and 0=I never feel this way. Min/max values: 0-60, with high scores indicating higher levels of social isolation. Scores at 6-months are reported.
Time Frame: 6 moths
Population: Only child reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 27.50 (6.08) | 28.24 (9.18) | 30.52 (9.93)

16. Secondary Outcome: Caregiver Mental Health (Caregiver Reports)
Description: Caregiver mental health functioning was assessed using 34-items from the Brief Symptom Inventory (BSI). The scale measures symptoms of anxiety, somatization and depression. Respondents were asked to rate how they felt emotionally, on a 5-point Likert scale, with 1=Never true, 2=rarely true, 3= true sometimes, 4= true most of the time and 5=always true. Min/max values: 34-170, with higher scores representing higher levels of caregiver mental distress. Scores at 6-months are reported.
Time Frame: 6 months
Population: Only caregiver reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 69.53 (26.71) | 65.88 (18.05) | 69.32 (19.81)

17. Secondary Outcome: Caregiver Parenting Stress (Caregiver Reports)
Description: Parenting stress was measured by 33 items from the Parenting Stress Index (PSI). The 33-item scale assesses symptoms related to parental distress, difficult child, and caregiver-child dysfunctional relationships. Respondents were asked to rate their parenting stress, on a 4-point Likert scale, with 1=strongly disagree, 2=somewhat disagree, 3=somewhat agree and 4=strongly agree. The theoretical range for this scale is 33-132, with high scores indicating high levels of parenting stress. Score at 6-months are reported.
Time Frame: 6 months
Population: Only caregiver reports were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Group-Cognitive Behavioral Therapy (G-CBT) | Multiple Family Group (MFG)
Number analyzed (Participants) | 28 | 25 | 31
score on a scale | 61.96 (12.99) | 62.52 (15.98) | 62.00 (13.44)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Usual Care: Children; Usual Care: Caregivers: Usual care consists of the traditional clinic intervention that focuses on testing services, ART treatment, and information about disease management.
- Group-Cognitive Behavioral Therapy (G-CBT): Children; Group-Cognitive Behavioral Therapy (G-CBT): Caregivers: Group Cognitive Behavioral Therapy (G-CBT): G-CBT consists of 10-session for HIV/AIDS-associated stigma, utilizing core components of CBT, including psychoeducation, cognitive restructuring, and skill-building to increase adaptive coping mechanisms.
- Multiple Family Group (MFG): Children; Multiple Family Group (MFG): Caregivers: Multiple Family Group (MFG): MFG consists of 10-sessions that strengthen family relationships intended to address HIV/AIDS-associated stigma at the individual level and within families. The core components of MFG are known as 4Rs and 2S's: rules, responsibility, relationships, respectful communication, stress and social support.
Arm/Group | Usual Care: Children | Group-Cognitive Behavioral Therapy (G-CBT): Children | Multiple Family Group (MFG): Children | Usual Care: Caregivers | Group-Cognitive Behavioral Therapy (G-CBT): Caregivers | Multiple Family Group (MFG): Caregivers
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26 | 1/34 | 1/29 | 0/26 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/34 | 0/29 | 0/26 | 0/34
Other Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/34 | 0/29 | 0/26 | 0/34

LIMITATIONS AND CAVEATS:
All study-related activities, including participant recruitment, data collection and intervention delivery, were conducted during the COVID-19 lockdown. The associated challenges may have impacted the study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT04528732/Prot_SAP_000.pdf